CLINICAL TRIAL: NCT07022938
Title: Efficacy and Safety of a Tablet Containing Palmitoyethanolamide, Alpha Lipoic Acid, Vitamin B12, Vitamin B6 , Vitamin B1, Nicotinamide, Magnesium, Zinc, Vitamin E, and Superoxide of Dismutase in Individuals Receiving Chemotherapy
Brief Title: Nutritional Supplement for Treating Chemotherapy Induced Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Prof. Triantafyllos Didangelos, Professor of Internal Medicine and Diabetology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2606/25.1.2021
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Neuropathy; Chemotherapy Induced Pain Neuropathy; Chemotherapy-Induced Peripheral Neuropathy
Keywords: cancer; neuropathy; chemotherapy induced neuropathy; supplement
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomised controlled placebo controlled study of a nutritional supplement intervention (epineuron) with 10 elements to investigate the effect in chemotherapy induced neuropathy
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epineuron (Active Comparator): Administration of a nutritional supplement with Palmitoylethanolamide (PEA, 300 mg), Superoxide Dismutase (SOD, 70 UI), Alpha Lipoic Acid (ALA, 300 mg), vitamins B6 (1.5 mg), B1 (1.1 mg), B12 (2.5 mcg), E (7.5 mg), Nicotinamide (9 mg) and minerals (Mg 30 mg, Zn 2.5 mg) in one tablet
  Interventions: Dietary Supplement: Epineuron
- Placebo (Placebo Comparator): similar tablet without active ingredients
  Interventions: Dietary Supplement: Placebo Tablets

INTERVENTIONS:
Dietary Supplement: Epineuron — Palmitoylethanolamide (PEA, 300 mg), Superoxide Dismutase (SOD, 70 UI), Alpha Lipoic Acid (ALA, 300 mg), vitamins B6 (1.5 mg), B1 (1.1 mg), B12 (2.5 mcg), E (7.5 mg), Nicotinamide (9 mg) and minerals (Mg 30 mg, Zn 2.5 mg) in one tablet
  Arms: Epineuron
Dietary Supplement: Placebo Tablets — placebo tablet without active ingredients
  Arms: Placebo

SUMMARY:
Administration of a nutritional supplement containing palmitoyethanolamide, alpha lipoic acid, vitamin B12, vitamin B6 , vitamin B1, nicotinamide, magnesium, zinc, vitamin E, and superoxide of dismutase in individuals receiving chemotherapy

DETAILED DESCRIPTION:
Investigation of effectiveness and safety of a nutritional supplement containing palmitoyethanolamide, alpha lipoic acid, vitamin B12, vitamin B6 , vitamin B1, nicotinamide, magnesium, zinc, vitamin E, and superoxide of dismutase in individuals receiving chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with cancer that have not received yet their treatment
* Patients that will be treated with platinum agents or taxanes

Exclusion Criteria:

* Not receiving dietary supplement
* Have already neuropathy
* Have already started chemotherapy
* Patients with uncontrolled diabetes

  -- Patients with chronic kidney disease
* Patiens with recent cardiovascular incident

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Neuropathic Pain Symptom Inventory | 6 months
  scale for neuropathic pain symptoms. A total intensity score can be calculated as the sum of the scores of the 10 descriptors. In addition, we propose to derive five subscores corresponding to the mean scores of the items belonging to each of the five factors identified in the factor analysis. three questions based on clinical examination to evaluate the intensity of pain evoked by brushing, pressure, cold or warm stimuli in the painful area on four-point categorical scales (absent, mild, moderate, severe). Clinical examination of evoked pain was standardized: tactile allodynia was evaluated with a soft brush (three movements), pressure allodynia was evoked by blunt pressure with a finger at a pressure that does not provoke pain in a normal area and glass tubes filled with hot (38-408C) or cold (22-248C) water were used to evaluate thermal allodynia.
PAIN Detect score | 6 months
  score for neuropathic pain, higher values indicate that the pain is neuropathic. A Pain DETECT score between-1 and 38 indicates the likelihood of a neuropathic pain component

SECONDARY OUTCOMES:
Visual Analogue scale | 6 months
  scale for pain , higher values indicate more severity of pain, scale 0-100
Nerve conduction velocity | 6months
  neurophysiological assessment of sural nerve
Vibration perception threshold | 6 months
  Vibration perception threshold was measured with biothesiometer

CONTACTS AND LOCATIONS:
Locations (1):
- University General Hospital of Thessaloniki AHEPA, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
Data privacy of participants